CLINICAL TRIAL: NCT04083066
Title: Open Randomized Prospective Clinical Study of Rituximab Combined With Fotemustine, Pemetrexed, Dexamethasone Versus Rituximab Plus Methotrexate, Cytarabine, and Dexamethasone in the Treatment of Primary Central Nervous System Lymphoma
Brief Title: Open Randomized Prospective Clinical Study of R-FPD Versus R-MAD Regimen in the Treatment of Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx20190221
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: rituximab; fotemustine; pemetrexed; ORR; OS; PFS
MeSH Terms: interventions — Rituximab; Methotrexate; Cytarabine; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rituximab combined with formoterol, pemetrexed, dexamethasone (Experimental): Rituximab 375mg/m2D0 is soluble in 0.9% NS, concentration 1mg/ml, micro pump is pumped for 4h Fotemustine 100mg/m2 D1 dissolved in 250mL 0.9% NS, intravenously for 1h, protected from light Pemetrexed 600mg/m2 D1 dissolved in 100ml 0.9% NS, intravenously 1h Dexamethasone 40mg D1-5 Dissolved in 100 ml 5% GS, intravenously (21 days is a cycle)
  Interventions: Drug: rituximab in combination with methotrexate, cytarabine and dexamethasone

INTERVENTIONS:
Drug: rituximab in combination with methotrexate, cytarabine and dexamethasone — Rituximab 375mg/m2D0 is soluble in 0.9% NS concentration 1mg/ml, micro pump is pumped in 4h HD-methotrexate 3.5g/m2 D1 dissolved in 0.9% NS intravenous drip HD-cytarabine 1g/m2 Q12H D2-3 Dissolved in 250ml 5% GS intravenously
  Dexamethasone 40mg D1-5 is dissolved in 100ml 5% GS intravenous drip (21 days is a cycle)

SUMMARY:
Comparison of the efficacy and safety of rituximab combined with fotemustine, pemetrexed, dexamethasone and rituximab in combination with methotrexate, cytarabine and dexamethasone as first-line regimens in the treatment of primary central nervous system lymphoma

DETAILED DESCRIPTION:
This is an open, randomized, prospective, multicenter clinical study designed to compare the efficacy and safety of R-FPD and R-MAD as first-line regimens in the treatment of primary central nervous system lymphoma. A total of 20 patients plan to participate in the study. The primary endpoints were objective response rate (ORR) and progression-free survival (PFS) and secondary endpoints including overall survival (OS), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

Age 14-75 years old; KPS score ≥ 60 points or ECOG score ≤ 2 points; expected survival period of more than 3 months; CD20 positive; PCNSL confirmed by tissue biopsy pathology (limited to brain, spinal cord, meninges and eyes, without lymphoma involving other parts of the body); no chemotherapy contraindications (blood and physiological examination results <7 days); At least one measurable lesion according to the RECIST criteria; There are no other serious diseases that conflict with this plan; There is a possibility of follow-up; When using other anti-tumor drugs at different times during this treatment, bisphosphonate anti-bone transfer therapy and other symptomatic treatments may be applied; Can understand the situation of this study and sign the informed consent form.

*: Pathological histology is subject to consultation by pathologists at provincial hospitals.

Exclusion Criteria:

Currently receiving other chemotherapy, radiotherapy and targeted therapy (chemotherapy within 3 weeks, radiotherapy within 2 weeks, or recovery from acute toxicity of any previous treatment); Pregnant or lactating women; There are any uncontrollable medical diseases (including active infection, uncontrolled diabetes, severe heart, liver, kidney dysfunction and interstitial pneumonia); combined with chemotherapy and other contraindications for chemotherapy; Those who have had other malignant tumors in the past; There are uncontrolled infected patients; Those who have a history of mental illness that is difficult to control; The investigator believes that it is not appropriate to participate in this test.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 months
  Objective Responder Rate
PFS | up to 24 months
  Progression Free Survival

SECONDARY OUTCOMES:
OS | up to 24 months
  Overall Survival
adverse events | up to 24 months
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi zhang, Dr., Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China